CLINICAL TRIAL: NCT07199920
Title: Implementation of New Multimodal MRI Sequences by Fingerprint to Improve Ischemic Stroke Examination, a Pilot Study and Proof of Concept
Brief Title: Implementation of New Multimodal MRI Sequences by Fingerprint to Improve Ischemic Stroke Examination.
Acronym: INDEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Grenoble Institut des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC23.0410
Record Dates: First submitted 2024-02-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Ischemic
Keywords: MRF (Magnetic Resonance Fingerprinting); stroke; MRI
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Every patient will perform classic brain MRI with additional MRF sequences.
  Interventions: Device: Achieva 3.0T dStream Philips

INTERVENTIONS:
Device: Achieva 3.0T dStream Philips — Classic and MRF sequences will be carried out on the clinical machine (Achieva 3.0T dStream Philips) of the IRMaGe platform (CHUGA, Université Grenoble Alpes, Inserm, CNRS).

SUMMARY:
Currently, standard brain MRI takes 20 to 25 minutes, but in the case of ischemic stroke, every minute counts to limit the extension of the necrotic core, with the possibility of recanalizing the occluded artery (intravenous thrombolysis and/or mechanical thrombectomy).

The recent concept of MRI "Fingerprint" (Magnetic Resonance Fingerprinting, MRF) allows the production of a rapid single sequence and the extraction of numerous parameters.

Demonstrating the feasibility and interpretability of multimodal MRI images acquired in MRF would make it possible to consider implementing and, ultimately, replacing conventional sequences, with the aim of shortening acute stroke management times, increasing the number of sequences acquired within a short timeframe (by increasing informativeness), and thus improving patients' short and long-term vital and functional prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Subacute ischemic stroke patients (< 15 days after onset)
* Middle cerebral artery or anterior cerebral artery territory stroke
* Modified Rankin Scale (mRS) = 0-4

Exclusion Criteria:

* MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Success rate and interpretability of images acquired in MRF | From enrollment to the end of the MRI exam
  Assessment of the success rate and interpretability (subjective evaluation with Likert scales of very satisfactory, satisfactory, insufficient, or unacceptable)

SECONDARY OUTCOMES:
Characterize and extract the physical parameters of the signal acquired with MRF. | From enrollment to the end of the MRI exam
  Comparison of MRF imaging metrics: signal-to-noise ratio (SNR) and contrast-to-noise ratio (CNR), using mean values per ROI (region of interest).
  Segmentation and comparison of lesions, with calculation of the Dice similarity coefficient and/or SSIM (Structural SIMilarity).
  Visualization and description of artifacts encountered during acquisition (e.g., motion).
  Quantification of delays:
  Acquisition time: retrieval of raw data directly from MRI consoles. Reconstruction time: measurement of computation times. Extraction of information on cerebral microvas

CONTACTS AND LOCATIONS:
Overall Officials: Loïc LEGRIS, Dr, Principal Investigator — llegris@chu-grenoble.fr
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No